CLINICAL TRIAL: NCT04475302
Title: Study to Evaluate the Effectiveness of BCG Vaccine in Reducing Morbidity and Mortality in Elderly Individuals in COVID-19 Hotspots in India
Brief Title: BCG Vaccine in Reducing Morbidity and Mortality in Elderly Individuals in COVID-19 Hotspots
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tuberculosis Research Centre, India (Other Government)
Collaborators: ICMR-National Institute for Research in Tuberculosis, Chennai, Tamil Nadu (Unknown); All India Institute of Medical Sciences (Other); National Institute for Research in Environmental Health, Bhopal, Madhya Pradesh (Unknown); National Institute of Occupational Health, Ahmedabad, Gujarat (Unknown); King Edward Memorial Hospital (Other); National Institute for Implementation Research on Non-Communicable Disease (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020010
Record Dates: First submitted 2020-07-16; First posted 2020-07-17 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: COVID
MeSH Terms: interventions — BCG Vaccine; Freeze Drying

STUDY DESIGN:
Intervention Model Description: In this study, as we are employing a control group that is not vaccinated against the disease to be prevented, but some clinical data are available to support the likely efficacy of the candidate vaccine, we will use unbalanced randomization and enrol participants to control group in the ratio of 2:1, so that majority of the study participant will receive the vaccine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): In the identified hotspots, BCG vaccine will be offered to all the elderly between 60 - 80 years of age. Those who get vaccinated will be followed for a period of 6-months.
  Interventions: Biological: BCG vaccine (Freeze-dried)
- Control arm (No Intervention): 1. in the hotspots, those who do not agree for vaccination, will be considered as controls. They will have an entry and exit interview at baseline and end of study period
  2. in situations where we are unable to enrol the required number of controls from the vaccination hotspot zones, then hotspots in the neighbouring area / wards where BCG is not offered will be taken as control sites. Elderly between 60-80 years in those areas would be considered as control sites for the study. The elderly participants will be approached for an entry and exit interview, if they agree. If they do not agree for an exit interview at the end of 6-months, then the status of those in the control group would be collected either from the corporation records / other medical database.

INTERVENTIONS:
Biological: BCG vaccine (Freeze-dried) — single dose of BCG vaccine (Freeze-dried) manufactured by Serum Institute of India, Pune. The composition of BCG vaccine is Live, attenuated BCG (Bacillus Calmette-Guerin Strain). (Each 1 ml contains between 2 x 106 and 8 x 106 Colony Forming Units (C.F.U.) with Diluent: Sodium Chloride Injection I.P.)
  Arms: Intervention arm

SUMMARY:
Rationale: SARS-CoV2 viral infection is spreading rapidly throughout the world and in India the epidemic poses a major threat to the public health system. Elderly individuals, especially those with diabetes, hypertension, other chronic diseases are at high risk of mortality. Strategies to protect these individuals are desperately needed to safeguard continuous patient care. Bacille Calmette-Guérin (BCG) is a vaccine against tuberculosis, with protective non-specific effects against other respiratory tract infections in in-vitro and in-vivo studies, and reported significant reductions in morbidity and mortality. Based on the capacity of BCG to reduce the incidence of respiratory tract infections in children and adults, to exert antiviral effects in experimental models; and to reduce viremia in an experimental human model of viral infection, the hypothesis is that BCG vaccination will partially protect against mortality in high-risk, elderly individuals.

Primary Objective: To evaluate the effectiveness of BCG vaccination in preventing morbidity and mortality due to COVID-19 in elderly individuals aged between 60 to 80 years living in COVID-19 hotspots in India.

Secondary objectives:

1. To evaluate the effectiveness of BCG vaccination in terms of

   1. reducing the cumulative incidence of hospital admission and Intensive Care admission
   2. reducing the incidence of other respiratory febrile illness
2. To determine the innate and adaptive immune responses, IgM, IgG and IgA antibody titers generated by BCG vaccination (both total and SARS-Cov2 specific) in a subset of individuals.
3. To measure biomarkers induced by BCG vaccination as correlates of risk/protection against SARS-Cov2 in a subset of individuals

Method and Analysis:

Study design: Intervention study Study population: Elderly 60 - 80 years of age residing in designated hotspots for SARS-Cov2 infection Study Intervention: One dose of 0.1ml BCG vaccine, given intradermally. Elderly individuals not vaccinated from the same hotspot area or from neighbouring hotspot wards areas will be considered as the controls. Study sites: Chennai, Mumbai, Ahmedabad, Bhopal, Jodhpur and New Delhi. Study Sample size: 1450 individuals between 60-80 years of age will receive BCG vaccination while 725 individuals will be controls without vaccination Study duration: 6 months/participant. Enrolment at each site will be over: 4 months. Each participant will be followed for 6 months post vaccination. Primary Outcome Measures: During the study period (6-months), Proportion of individuals receiving the BCG vaccination who are asymptomatic but become PCR-positive or seroconvert during the 6-month of study period. Proportion of patients with development of COVID-19 disease (either PCR-positive or seroconvert with symptoms) during the study period. Proportion of patients with Severe COVID-19 disease and death due to Covid-19 disease

DETAILED DESCRIPTION:
Recruitment area: Under the Lockdown 2.0, the country has been classified into three key zones-Red, Orange and Green (26). These zones will support the cluster containment plan announced by the government, while opening up the rest of the places.

Green Zone: Places which have so far not reported even a single COVID-19 positive case will be declared as Green Zone under Government's new plan. This means nearly 400+ districts of India might qualify to be tagged as Green Zone.

Orange Zone: Orange zone may see opening of limited public transport and also allow exemptions for essential services personnel and farming and harvest activity for the ongoing season. Orange zone will have less than 15 cases of COVID-19.

Red Zone: A district or cluster declared as a red zone, will see severe restrictions with zero or no activity allowed. Typical understanding is that any place with more than 15 COVID-19 positive cases can be declared as a red zone. Investigators will include the Red & Orange zones of Delhi, Madhya Pradesh, Maharashtra, Gujarat, Tamilnadu, Rajasthan and other interested states for this study.

Recruitment methods: Participants would be recruited through (i) information presented in community organizations, hospitals, colleges and other institutions to the general public. (ii) From a line list prepared of adults above the age of 60 years from Census data for the hotspot areas. (iii) Participants will also be recruited by use of an advertisement +/- registration form formally approved by the ethics committee(s) and distributed or posted in the

1. newspapers or other literature for circulation.
2. Via presentations (e.g. presentations at lectures or invited seminars). (iv) Community Advisory Board will be created for this study and help of the members of this board will be taken for recruitment to the study Interested individuals will be provided detailed information about the study and the requirements for participation will be provided. Participants will be given brochure about the study and patient information sheet. They will have the opportunity to ask any questions they might have and to talk to a study team member. If they are still interested and willing to participate, they will be invited to participate in screening evaluation procedure.

Study Procedures: Participants meeting inclusion criteria will be recruited in a nonrandomized manner after obtaining their consent to participate to the study. An information document that clearly indicates the risks and the benefits associated with the participation to the study will be given to each patient before signing consent. Regarding participant identification, a study number will be assigned sequentially to included participants, according to the range of patient numbers allocated to each study center.

Participants will be seen at baseline for enrolment, initial data collection (a detailed medical history including h/o previous BCG vaccination and evidence of BCG vaccination scar to be noted), Chest x-ray PA view to rule out PTB, blood sampling for antibody testing (2 ml) and PCR (nasopharyngeal swab).

Eligible participants will be administered BCG at day 0. Participants will be followed up weekly by phone for first 2 months and asked to complete a standardized questionnaire. Month 1, 3 & 6 will be visit in person while Month 2 & 5 will be completed over phone. Participants would be tested for COVID antibodies at month 3 and month 6. If positive, nasal/throat swab would be collected for PCR testing for confirmation. Participants will also be asked to call the study staff in the event of any adverse reactions or illness. Participants will thereafter be followed up monthly for six months.

Participants will be given a diary card (paper), with instructions to fill in case of adverse events, along with the emergency 24 hour telephone number to contact the on-call study physician if needed. They will be instructed on how to self-assess the severity of these AEs. There will also be space on the diary card to self-document unsolicited AEs, and whether medication was taken to relieve the symptoms.

In addition to blood, nasopharyngeal swabs will be collected from all participants.

qRT- PCR test will be considered to reconfirm the qRT-PCR positive / negative status at enrolment. In a subset of this cohort (15% of the sample), consenting for immunological substudy, 20 ml of blood will be collected at baseline for immunological and biomarker analysis. They will also provide additional blood samples (20 ml) at 1, 3 and 6 months post vaccination for immunological and biomarker studies.

Blood collection: Investigators will collect 2 ml of venous blood after obtaining consent from participants. Investigators will collect the specimen using a syringe following all the safety precautions and transfer the specimen to serum separator tubes. After completion of sample collection from all eligible participants, the specimen will be transported to the nearest District Public Health Laboratory (DPHL)/Virus Research and Diagnostic Laboratory Network (VRDLN) laboratory in cold chain. In the laboratory, serum will be separated and used for rapid antibody testing. Detection of SARS-CoV 2 specific antibodies will be performed using a ICMR validated SARS-CoV-2 Antibody Test. The Lateral Flow-based immune-chromatographic test detects SARS-CoV 2 specific antibodies (IgG/IgM) with a turnaround time of 15-20 mins. Presence of coloured bands at Test and Control lines will indicate the presence of SARS-CoV-2 antibodies (positive result) in the specimen. Absence of coloured band in Test line will indicate the absence of SARS-CoV-2 antibodies (negative result).

Immunology analysis: The primary variables of interest of immune response to vaccines will be the percentage of CD4+ and CD8+ T cells that express IFN-γ, TNF, IL-2, IL-17, IL-22, CD107a, Perforin, Granzyme B and Granulysin alone or in combination in response to stimulation with SARS-Cov-2 and BCG antigens. Secondary variables of interest would be the response of trained monocytes and other innate immune cells including NK cells, NKT cells, gd T cells and MAIT cells. Response will be measured by flow cytometry in the intracellular cytokine staining (ICS) assay. Blood collected for immunological studies will be utilized as follows: PBMC isolation and storage for immunology studies described above; Whole blood in Lithium Heparin microtainer for absolute blood cell counting by flow cytometry (deconvolution for transcriptomics) and for Interferon Gamma Release Assays; plasma and serum for soluble immune mediators by ELISA and for total and SARS-Cov2 specific IgG, IgM and IgA ELISA.

Diagnostic tests:

PCR: Molecular diagnosis of SARS-Cov2 will be done by using RT-PCR kits according the ICMR guidelines. Serology: Antibody IgG/IgM Covid-19 rapid test kit will be used. Chest x-ray along with symptom screening: To rule out tuberculosis

Subgroup Analysis

1. The primary analysis will be performed using the whole cohort
2. A stratified analysis will be undertaken for various age groups and by risk groups based on co-morbidity. This will allow vaccine effectiveness to be assess in more homogeneous subgroups and to check for effect of modification across strata
3. Stratified analysis will also be done for various geographic distribution and occupation
4. Immunological analysis will be carried out in a subset of individuals (n=200)

ELIGIBILITY:
Inclusion Criteria:

* Adults 60 years of age or older (<100 years) with general good health, as confirmed by history and physical examination.
* No known history of HIV or on immunosuppressive drugs for malignancy or transplant
* Provide a signed and dated informed consent form

Exclusion Criteria:

* Positive for SARS-Cov2 infection
* Known HIV or other immune-suppressive treatments for malignancy or transplant
* Recently diagnosed as TB or currently on anti-TB treatment or anti-psychiatric medications
* Has any BCG vaccine contraindication
* H/o of previous administration of experimental MTB vaccines within the past 6 months.
* Sick and moribund individuals with Karnofsky score <50

  * Elderly individuals with or without co-morbid conditions like Diabetes mellitus, or Hypertension or Hyperlipidemia will be considered for this study, if they are on regular treatment.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2175 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Mortality due to COVID-19 disease | 6 months from study start date
  Number of deaths due to COVID-19 disease

SECONDARY OUTCOMES:
Hospital admission and ICU admission due to Covid-19, Severity of Covid-19 (mild, moderate or severe), Hospital admission due to other respiratory febrile illness, immunological outcomes in the sub study | 10 months from study start date
  Number of hospital admissions and ICU admissions due to Covid-19 and other respiratory disease, Number of COVID-19 cases reported based on severity level (mild, moderate or severe) and immunological outcomes in the sub study (baseline and at 1, 3 and 6 months post vaccination).

CONTACTS AND LOCATIONS:
Overall Officials: Padmapriyadarsini Chandrasekaran, MBBS,DNB,MS, Principal Investigator — National Institute for Research in Tuberculosis; Anant Mohan, Principal Investigator — All India Institute of Medical Sciences; Randeep Guleria, Principal Investigator — All India Institute of Medical Sciences; Tiwari R R., Principal Investigator — National Institute for Research in Environmental Health; Yogesh Sabde, Principal Investigator — National Institute for Research in Environmental Health; Kamalesh Sarkar, Principal Investigator — National Institute of Occupational Health; Asha Keetharam, Principal Investigator — National Institute of Occupational Health; Hemant Deshmukh, Principal Investigator — KEM Hospital; Rujuta Hadaye, Principal Investigator — GSMC and KEM Hospital; Toteja G.S., Principal Investigator — National Institute for Implementation Research on Non-Communicable Disease; Subash Babu, MBBS, PhD, Principal Investigator — NIH-International Center for Excellence in Research
Locations (1):
- Tuberculosis Research Centre, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No